CLINICAL TRIAL: NCT02542956
Title: Prospective, Randomized, Controlled Comparison of Local Anesthetic Infusion Pump Versus DepoFoam Bupivacaine For Pain Management After Abdominoplasty and TRAM Flap Breast Reconstruction.
Brief Title: Comparison of Local Anesthetic Infusion Pump Versus DepoFoam Bupivacaine for Pain Management
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Donna Tepper M.D, Plastic Surgeon, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SR91333
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Pain
Keywords: Tummy tuck (abdominoplasty); Breast Surgery
MeSH Terms: conditions — Pain | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exparel (Active Comparator): Injection of Exparel
  Interventions: Drug: Exparel
- Marcaine (Active Comparator): Receive Marcaine in a pain pump or by injection
  Interventions: Drug: Marcaine

INTERVENTIONS:
Drug: Exparel — receive Exparel by injection
  Arms: Exparel
Drug: Marcaine — receive Marcaine in a pain pump
  Arms: Marcaine
Drug: Marcaine — receive Marcaine by injection
  Arms: Marcaine

SUMMARY:
The purpose of this study is to identify the best pain management for patients undergoing abdominoplasty after massive weight loss or transverse rectus abdominis myocutaneous (TRAM) flap for breast reconstruction. The investigator is conducting this study to compare the effectiveness of a continuous infusion pain pump versus a locally injectable long-acting anesthesia (DepoFoam bupivacaine) versus standard injectable anesthesia (bupivacaine) for post surgical pain control. These drugs and devices are approved by the FDA (Food and Drug Administration) for the purpose of pain control after surgery, and have been used for this purpose before.

DETAILED DESCRIPTION:
The purpose of this study is to identify the best pain management for patients undergoing abdominoplasty after massive weight loss or transverse rectus abdominis myocutaneous (TRAM) flap for breast reconstruction. The investigator is conducting this study to compare the effectiveness of a continuous infusion pain pump versus a locally injectable long-acting anesthesia (DepoFoam bupivacaine) versus standard injectable anesthesia (bupivacaine) for post surgical pain control. These drugs and devices are approved by the FDA (Food and Drug Administration) for the purpose of pain control after surgery, and have been used for this purpose before.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing abdominoplasty or TRAM flap breast reconstruction

Exclusion Criteria:

* A medical condition that could interfere with study participation
* Body weight less than 50 kg
* Participating in another study involving an investigational medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Recurrence of Pain | 30 minute to 72 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Donna Tepper, M.D, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States